CLINICAL TRIAL: NCT01434888
Title: A Phase I, Randomized, Double-masked, 3-period Cross-over Clinical Study to Compare the Pharmacokinetics, Safety and Tolerability of the Preservative-free Fixed Dose Combination of Tafluprost 0.0015% and Timolol 0.5% Eye Drops to Those of Preservative-free Tafluprost 0.0015% and Timolol 0.5% Eye Drops in Healthy Volunteers
Brief Title: Pharmacokinetics, Safety and Tolerability of the Preservative-free Fixed Dose Combination of Tafluprost 0.0015% and Timolol 0.5% Eye Drops
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santen Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 201150; 2011-001778-24 (EudraCT Number)
Record Dates: First submitted 2011-09-12; First posted 2011-09-15 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Volunteers
Keywords: pharmacokinetics
MeSH Terms: interventions — Ophthalmic Solutions; Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tafluprost 0.0015% (Active Comparator)
  Interventions: Drug: Preservative free tafluprost 0.0015% eye drops
- Timolol 0.5% (Active Comparator)
  Interventions: Drug: Preservative free timolol 0.5% eye drops
- Fixed-dose combination of tafluprost 0.0015% and timolol 0.5% (Experimental)
  Interventions: Drug: Preservative free FDC of tafluprost 0.0015% and timolol 0.5% eye drops

INTERVENTIONS:
Drug: Preservative free tafluprost 0.0015% eye drops — Preservative free tafluprost eye drops will be administered once daily at 09:00 into both eyes for seven days. For masking purposes vehicle eye drops will be administered in the evening at 21:00.
  Arms: Tafluprost 0.0015%
Drug: Preservative free timolol 0.5% eye drops — Preservative free timolol eye drops will be administered into both eyes twice daily at 9:00 and 21:00 for seven days
  Arms: Timolol 0.5%
Drug: Preservative free FDC of tafluprost 0.0015% and timolol 0.5% eye drops — Preservative free fixed-dose combination eye drops will be administered into both eyes once daily at 9:00 for seven days. For masking purposes vehicle eye drops will be administered in the evening at 21:00.
  Arms: Fixed-dose combination of tafluprost 0.0015% and timolol 0.5%

SUMMARY:
The objective of this study is to investigate the pharmacokinetics, safety and tolerability of the preservative-free fixed-dose combination of tafluprost 0.0015% and timolol 0.5% (FDC) to those of preservative-free tafluprost 0.0015% and timolol 0.5% eye drops in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 45 years
* Good general health
* Meet best corrected ETDRS visual acuity

Exclusion Criteria:

* Significant systemic or ocular disease
* History of eye surgery, including refractive surgery
* Allergy or hypersensitivity to study drug
* Low heart rate (<50 bpm)
* Clinically relevant low blood pressure
* Asthma
* Bradycardia
* Use of contact lenses within one week prior to screening or during the study
* Clinically significant obesity (body mass index > 30 kg/m2)
* Blood donation within 2 months prior to screening
* Females who are pregnant or lactating and females not using adequate contraceptives

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics after single and repeated administration of preservative-free FDC, tafluprost and timolol eye drops. | There are 3 cross-over treatment periods, plasma concentrations will be measured on Day 1 and Day 7
  The primary evaluation of pharmacokinetics will be based on the plasma concentration of tafluprost acid and timolol.

SECONDARY OUTCOMES:
Safety and tolerability after single and repeated administration of preservative-free FDC, tafluprost and timolol eye drops. | Day 1 and Day 7 of treatment periods I, II and III.
  The changes from screening/baseline will be evaluated in following variables:visual acuity, IOP, biomicroscopy and ophthalmoscopy findings and drop discomfort.
  Adverse events will be followed from screening to post-study visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital Eye Clinic, Kuopio, Finland